CLINICAL TRIAL: NCT00503295
Title: A Phase 2 Study of Intravenous REOLYSIN® (Wild-Type Reovirus) in the Treatment of Patients With Bone and Soft Tissue Sarcomas Metastatic to the Lung
Brief Title: Safety and Efficacy Study of REOLYSIN® in the Treatment of Bone and Soft Tissue Sarcomas Metastatic to the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 014
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2012-05

CONDITIONS: Osteosarcoma; Ewing Sarcoma Family Tumors; Malignant Fibrous Histiocytoma; Sarcoma, Synovial; Fibrosarcoma; Leiomyosarcoma
Keywords: reovirus; oncolytic virus; sarcoma; REOLYSIN; Oncolytics Biotech
MeSH Terms: conditions — Osteosarcoma; Histiocytoma, Malignant Fibrous; Sarcoma, Synovial; Fibrosarcoma; Leiomyosarcoma; Sarcoma | interventions — reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: REOLYSIN® — REOLYSIN® is given intravenously at a dose of 3x10E10 TCID50 over 60 minutes on Days 1-5 of a 28 day cycle.

SUMMARY:
The purpose of this Phase 2 study is to investigate whether intravenous administration of REOLYSIN® therapeutic reovirus is safe and effective in the treatment of patients with bone and soft tissue sarcomas metastatic to the lung.

DETAILED DESCRIPTION:
Sarcomas are uncommon mesenchymal malignancies that encompass a variety of tumors of soft tissue or bone. Included in this study are patients with osteosarcoma, Ewing sarcoma family tumors, malignant fibrous histiocytoma, synovial sarcoma, leiomyosarcoma and fibrosarcoma. Patients with these lesions presenting with metastatic disease remain largely incurable. In all sarcomas, the lungs are by far the most frequent site of metastases.

There is a need for new therapies that have activity against these types of sarcomas. REOLYSIN® is an unmodified oncolytic reovirus which replicates selectively in ras transformed cells causing cell lysis. Activating mutations in ras or mutations in oncogenes signaling through the ras pathway may occur in as many as 80% of human tumors. Such mutations have been described in many of the common sarcomas of childhood and adults. REOLYSIN® demonstrated excellent anti-tumor activity in vitro and in vivo in childhood sarcoma cell lines.

Further supporting the development of REOLYSIN® in the context of sarcomas as detailed in this study, is the fact that sarcomas resistant or refractory to conventional chemotherapy may remain clinically responsive to viral therapy. Sarcoma patients with pulmonary metastases may be especially suitable for studies with REOLYSIN® due to rapid selective uptake of the virus by the lungs.

This Phase 2 study is designed to characterize the efficacy and safety of REOLYSIN® given intravenously over 5 days every 4 weeks in patients with bone and soft tissue sarcomas metastatic to the lung. Safety data, including laboratory parameters and adverse events, will be collected for all patients in order to determine the toxicity and reversibility of toxicity of REOLYSIN® therapy. Response will be assessed using radiographic imaging every 2 cycles of therapy.

OBJECTIVES:

1. To measure tumor responses and duration of response, and describe any evidence of antitumor activity of intravenous multiple dose REOLYSIN® in patients with bone and soft tissue sarcomas metastatic to the lung.
2. To evaluate safety of intravenous multiple dose REOLYSIN®.

ELIGIBILITY:
Inclusion Criteria:

* have a bone or soft tissue sarcoma metastatic to the lung deemed by a physician to be unresponsive to, or untreatable by, standard therapies. Acceptable histologies include only osteosarcoma, Ewing sarcoma family tumors, malignant fibrous histiocytoma, synovial sarcoma, fibrosarcoma and leiomyosarcoma
* have ≥ 2 measurable lesions in the lungs detectable on CT scan
* all residual adverse effects related to any prior anti-cancer therapy including, but not limited to, chemotherapy, biologic therapy, radiotherapy or surgical procedures must have resolved to Grade 1 or lower (as defined by the Common Terminology Criteria for Adverse Events, Version 3.0) before study therapy is initiated
* have received NO chemotherapy, radiotherapy, immunotherapy, hormonotherapy or surgery (except skin surgeries and minor biopsies) within 28 days prior to receiving REOLYSIN®
* have ECOG Performance Score of ≤ 2
* have life expectancy of at least 3 months
* Absolute neutrophils ≥ 1.5 x10^9/L; hemoglobin ≥ 9.0g/dL; platelets ≥ 100 x 10^9/L
* SGOT/SGPT (AST/ALT) ≤ 2.5 x ULN; bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN
* negative pregnancy test for females of childbearing potential

Exclusion Criteria:

* have inadequate pulmonary function defined as a forced expiratory volume in 1 second (FEV1) less than 50% of predicted
* be on immunosuppressive therapy; have known HIV infection or active hepatitis B or C
* have clinically significant pulmonary or cardiac disease
* have dementia or altered mental status that would prohibit informed consent
* have any other severe or acute chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgement of the Principal Investigator, would make the patient inappropriate for this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-06; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) and partial response (PR) as well as prolonged stabilization of disease (SD) will be considered indicative of response. RECIST criteria will be utilized to assess radiographic response. | For PR or CR, changes in tumor measurements must be confirmed 4 weeks after the criteria for response are first met. For SD, follow-up measurements must have met the SD criteria at least once after trial entry at a minimum interval of 12 weeks.

SECONDARY OUTCOMES:
Safety data, including laboratory parameters and adverse events, will be collected for all patients in order to determine the qualitative and quantitative toxicity, and reversibility of toxicity, of REOLYSIN®. | within 30 days of the last dose of REOLYSIN®

CONTACTS AND LOCATIONS:
Overall Officials: Karl Mettinger, MD, PhD, Study Director — Oncolytics Biotech
Locations (4):
- United States (4):
  - University of Michigan Medical School, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Montefiore Medical Center/Albert Einstein College of Medicine, The Bronx, New York
  - Institute of Drug Development, Cancer Therapy Research Center, San Antonio, Texas

REFERENCES:
- See also: Click here for more information about this study: Clinical Trials - Phase II Sarcomas Trial - United States — http://oncolytics.ca/clinical-trials/12